CLINICAL TRIAL: NCT06520085
Title: Optimizing Recovery After Reverse Shoulder Arthroplasty With a Personalized Mobile Health Application
Acronym: TRAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Anna ziekenhuis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAPP; N22.075 (Other: METC Maxima Medical Centre, Eindhoven-Veldhoven)
Record Dates: First submitted 2024-07-05; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Osteoarthritis
Keywords: Reverse Shoulder Arthroplasty; mHealth; Perioperative Care; Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study is a multicentre, single-blinded (assessor), two-armed, parallel-group RCT designed to evaluate the effectiveness of a an interactive mHealth application to standard care (non-interactive app) in the rehabilitation period of patients undergoing RSA.
Who Masked: Outcomes Assessor
Masking Description: Because the application relies on interaction between patient and clinical care team, both the patient and clinicians cannot be blinded. The researcher that will perform data analysis will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized rehabilitation program (Experimental): The intervention group receives an interactive app that is different from the control is different from the control group in that it provides interactive and personalized information and a personalized rehabilitation program. Both the timing and the amount and nature of the exercises are personalized.
  Interventions: Other: interactive mHealth application for patients undergoing RSA
- Standard care (Active Comparator): The control group will receive postoperative information and a rehabilitation program via the non-interactive application, which is current standard care
  Interventions: Other: interactive mHealth application for patients undergoing RSA

INTERVENTIONS:
Other: interactive mHealth application for patients undergoing RSA — Patients will receive interactive information via an mHealth application tailored to their needs and progress during the rehabilitation period after RSA.

SUMMARY:
Background: Mobile health (mHealth) - the use of medical applications in healthcare settings - include tools that can support self-management after surgery and thereby contribute to early postoperative recovery. Providing patients with timely and interactive information through mHealth is hypothesized to positively influence recovery after reverse shoulder arthroplasty (RSA).

Aim: The aim of this study is to determine the effectiveness of interactive and personalized information and rehabilitation protocol with a mobile application compared to generic information and generic rehabilitation protocol (standard care) on postoperative recovery in patients undergoing primary RSA.

Methods and analysis: A multicentre randomised controlled trial will be conducted in two Dutch hospitals. In total 170 patients undergoing elective, primary RSA will be included. Participants will be randomly allocated to one of the two groups on a 1:1 ratio. The intervention group will receive interactive postoperative information on a daily basis. The control group will receive standard care. The primary outcome is defined as functional recovery measured using the Oxford Shoulder Score (OSS) at 6 weeks. Secondary outcomes are: pain, physical functioning, quality of life, length of stay, complications, treatment satisfaction and app use. The between group difference will be analysed using linear mixed-effects regression.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing elective reverse shoulder arthroplasty

Exclusion Criteria:

1) do not own or are not able to operate a smart device; 2) are scheduled for revision surgery; 3) have a fracture as primary diagnosis; 4) an additional muscle transfer needs to be performed; or 5) are unable to read and understand the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative shoulder functioning | bssix weeks, three months and 1 year
  Shoulder functioning measured with the Oxford Shoulder Score

SECONDARY OUTCOMES:
Shoulder pain | baseline, daily during the first 6 weeks, 3 months and 1 year
  Shoulder pain measured using the Numeric Rating Scale
Shoulder disability | baseline, six weeks, three months and 1 year
  shoulder disability measured using the Disability of the Arm, Shoulder and Hand
Range of Motion of the Shoulder | baseline, six weeks, three months and 1 year
  Range of Motion of the Shoulder measured with the goniometer
Satisfaction with the Application | six weeks, three months and 1 year
  Satisfaction with the Application measured with a five-point likert scale
Readmission rate | 1 year
  Readmission rate related to RSA
Complication rate | 1 year
  Complication rate related to RSA

CONTACTS AND LOCATIONS:
Locations (1):
- VieCuri Medisch Centrum, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD may be requested through the contact person. Upon reasonable request these may be provided on a case by case basis.

REFERENCES:
- [Derived] Crutsen JRW, Heerspink FOL, Kornuijt A, Ascencio J, van der Weegen W, Timmers T, Craamer C, van Raay JJAM, Hollman F, Janssen ERC. Optimizing recovery after reverse shoulder arthroplasty with a personalised mobile health application compared to generic digital information: a protocol of a multicentre randomised controlled trial. BMC Musculoskelet Disord. 2025 Jul 4;26(1):642. doi: 10.1186/s12891-025-08857-9. PMID 40616068